CLINICAL TRIAL: NCT02431936
Title: Effectiveness of Prazosin on the Urinary Sodium Excretion Response to Mental Stress in a Randomized Double Blind Placebo Controlled Design
Brief Title: Effectiveness of Prazosin on the Urinary Sodium Excretion Response to Mental Stress
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Augusta University (Other)
Collaborators: The University of Texas at Arlington (Other)
Responsible Party: Principal Investigator, Gregory Harshfield, Director, Augusta University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 611851
Record Dates: First submitted 2015-04-28; First posted 2015-05-01 (Estimated); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Hypertension; Stress, Psychological; Blood Pressure
Keywords: Stress; Blood Pressure; Salt Sensitivity; Renin-Angiotensin-Aldosterone System; Sympathetic Nervous System
MeSH Terms: conditions — Hypertension; Stress, Psychological | interventions — Prazosin; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prazosin (Experimental): Prescription for 1mg oral Prazosin twice per day will be administered for 71/2 days.
  Interventions: Drug: Prazosin
- Placebo (Placebo Comparator): Prescription for placebo identical to Prazosin dosage will be administered for twice daily for 71/2 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prazosin — Double blind placebo controlled cross over trial to determine effectiveness of alpha adrenergic blocker in reducing sodium retention during stress.
  Other Names: minipress
  Arms: Prazosin
Drug: Placebo — Sugar pill made to look identical to Prazosin intervention.
  Other Names: sugar pill
  Arms: Placebo

SUMMARY:
High blood pressure, or hypertension, is a serious problem in the African-American (AA) population which affects nearly 7 of every 10 AAs in our area. Previously the investigators showed that a significant number of AAs held onto or retained salt during mental stress (sodium retainers). The investigators believe that the increased salt load and resulting blood pressure load contributes to the eventual development of hypertension in these individuals. The purpose of this study is to find out if this response is due to the direct stimulation of the kidney (the organ that controls salt levels in the body, by the brain). To do this, the investigators will determine if a drug that stops the connection between the brain and the kidney during mental stress will prevent sodium retention in sodium retainers. Prazosin is an alpha adrenergic receptor blocker that has been approved by the Food and Drug Administration (FDA). None of the subjects who participate in this study have high blood pressure. The subjects will not know which testing week is the drug week and which is the placebo week.

DETAILED DESCRIPTION:
High blood pressure, or hypertension, is a serious problem in the African-American (AA) population which affects nearly 7 of every 10 AAs in our area. Previously the investigators showed that a significant number of AAs held onto or retained salt during mental stress (sodium retainers). The investigators believe that the increased salt load and resulting blood pressure load contributes to the eventual development of hypertension in these individuals. The purpose of this study is to find out if this response is due to the direct stimulation of the kidney (the organ that controls salt levels in the body, by the brain). To do this, the investigators will determine if a drug that stops the connection between the brain and the kidney during mental stress will prevent sodium retention in sodium retainers. Prazosin is an alpha adrenergic receptor blocker that has been approved by the Food and Drug Administration (FDA). None of the subjects who participate in this study have high blood pressure. The subjects will not know which testing week is the drug week and which is the placebo week. Participants will test twice during this study, one of the weeks they will take Prazosin daily and the other week of testing they will take a placebo (sugar pill) daily in order to see if Prazosin changes how their body handles salt during stress. The participants will not be informed as to which of the testing weeks is the Prazosin week or the placebo week. This study will involve a screening visit, two first dose visits and two testing weeks over an approximate 5 week period (this include a one week "washout" period). Each testing week will have a 3 day salt-controlled diet prior to testing and an approximate 3-hour testing period on Day 4. The 3-hour testing period will include 10 minutes of a baseline rest, 45 minutes of mild stress (competitive video game), and 45 minutes of a recovery rest. A total of 4 blood and 4 urine samples will be collected during the 3-hour period. Each blood draw will consist of about 4 teaspoons for a total of 16 teaspoons. If the participants are female, a pregnancy test will be performed at the beginning of each testing visit (screening, first dose-1, test day-1, first dose-2 and test day-2) to confirm that they are not pregnant. Muscle sympathetic nerve activity will be measured during testing through the insertion of electrodes just below the knee on the outer part of the right leg. Additionally, an IV infusion will be administered for the phenylephrine challenge to insure total blockade of the sympathetic nervous system.

ELIGIBILITY:
Inclusion Criteria:

* of good general health
* not on any prescription medications
* between the ages of 18 and 50 years
* not pregnant
* African-American male or female

Exclusion Criteria:

* not African-American
* pregnant
* taking medications that will affect blood pressure
* not in good general health
* younger than 18 years of age or older than 50 years of age

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2015-04; Primary Completion 2019-04-16 (Actual); Study Completion 2019-04-16 (Actual)

PRIMARY OUTCOMES:
Urinary sodium excretion rate | 2 hours
  Primary variable of interest is the difference in stress induced changes in sodium excretion between placebo and treatment conditions in African-Americans who retain sodium during stress.

SECONDARY OUTCOMES:
Hemodynamics: change in systolic blood pressure | 2 hours
  Measures of change in systolic blood pressure compared to changes in sodium excretion in treatment versus placebo in African-Americans who retain sodium during stress.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A Harshfield, PhD, Study Director — Augusta University
Locations (1):
- Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Dissemination will be carried out in a variety of ways that will be accessible to other scientists studying psychosocial stress, hypertension, and the control of fluid-electrolyte balance and blood pressure. These include publications made available through PubMed-cited journals and presentations at scientific meetings and various organizations.
Supporting Information: Study Protocol